CLINICAL TRIAL: NCT04784364
Title: Biologics and Clinical Immunology Cohort At Sinai
Acronym: BACICS
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Rachel Miller, Chief, Division of Clinical Immunology, Icahn School of Medicine at Mount Sinai
Other Study IDs: HSM 20-01252
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Immunological Disease; Autoimmune Diseases; Primary Immune Deficiency
Keywords: Asthma; Immune Deficiency; Autoimmunity
MeSH Terms: conditions — Immune System Diseases; Autoimmune Diseases; Primary Immunodeficiency Diseases; Asthma; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Plasma blood, Peripheral blood mononuclear cells (PBMC), Salivary DNA self-collection, Buccal swabs, Tape strips on skin, Nasopharyngeal swab for nasal epithelial cell, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study team plans to establish a bioregistry of patients receiving biologic therapy as part of their standard treatment at the Mount Sinai Therapeutic Infusion Center and affiliated practices. The study team will to apply state-of-the-art approaches to assessing and predicting immunological and clinical responses associated with these standards and prescribed treatments. The approach is twofold. The first component is to establish a robust and flexible biorepository and database that includes demographic, immunologic, exposure and clinical records, and can facilitate research across disciplines, and across other registries affiliated with Mount Sinai. The second component is to address specific key research questions focused on using novel diagnostics to increase the effectiveness of biologic treatment. Most patients will be recruited from the Mount Sinai Therapeutic Infusion Center (TIC), although others receiving infusions elsewhere or at home will be recruited from outpatient Sinai affiliated clinical practices.

DETAILED DESCRIPTION:
The study team proposes a twofold approach to determine how immunophenotype may affect the course of clinical immunological disease for patients receiving biologic therapy. First, the team intends to establish a biorepository and database that includes demographic, immunologic, exposure and clinical records. The registry will be set up to facilitate research across disease disciplines, and across other registries affiliated with ISMMS. Second, over time, the team aims to address specific and an increasing number of research questions focused on using novel diagnostics to increase the effectiveness of biologic treatment as outlined below. Most subjects will be recruited from the Mount Sinai Therapeutic Infusion Center (TIC), although others receiving infusions elsewhere or at home will be recruited from outpatient affiliated clinical practices during scheduled medical visits.

Specific Aims:

1. (Overarching) Build a repository of biological specimens, questionnaire data, and apply state-of-the-art assessment tools to assess the current immunological and clinical condition, and changes over time. Specimens and data will be collected in a manner that can readily incorporate new technology, new research questions, link to intelligent analytics, and provide a resource for future consortia across disciplines. An infrastructure will be created that includes a multi-disciplinary Steering Committee to facilitate spinoff research studies and harmonize protocols within the TIC and across the Sinai system, resolve procedural questions, and communicate updated policies to referring physicians.

Additional initial specific scientific aims related to responses to biologics prescribed as part of standard practice that will be considered in this proposal are to determine:

2 . Effects of anti-IgE therapy on IgE phenotypes, maturation and production, and clinical outcomes.

3. Effects of anti-IgE and anti-IL-5 therapies on dopaminergeric pathways and clinical outcomes.

4. Effects of anti-TNF, anti-CD20, and other biologic therapies on immunological and clinical outcomes.

5. Effects of IVIG therapy on immunological and clinical course in Common Variable Immune Deficiency.

Futures studies will focus on Clinical Decision Support (CDS), Artificial Intelligence, and use of technology to inform and educate current TIC patients. Future studies also will feature studies related to immunological and clinical responses to additional biological therapies.

Background The prescription of biological agents and immune modulators to treat chronic immunological-based diseases continues to expand. This trend is predicted to continue. Applying data-driven and immunophenotype-driven approaches to their use could reveal additional pharmacologic targets and signal disease presence or relapse prior to the onset of clinical symptoms. These advances in precision medicine also may reduce adverse drug reactions and help control overall cost of healthcare associated with inefficient and 'trial and error' prescribing. They also may provide information on susceptible individuals and their appropriate care during healthcare crises, such as the current COVID-19 pandemic.

Despite these developments, prospective studies and clinical trials that feature immunophenotyping to facilitate 'real world' therapeutic decision-making are limited. More comprehensive immunophenotyping has predicted clinical responses to cancer immunotherapy, suggesting that this approach may translate to immunologically-mediated nonmalignant diseases. But widespread application to multiple chronic diseases is limited by several research gaps. These include determination of: 1) new biomarkers (discovery, validation) that may inform clinicians of drug responsive endotypes, 2) biomarkers that predict disease course over time in replicate studies, 3) optimal methods to link immunophenotype with analytic diagnostic and clinical decision-making tools to predict disease course, 4) factors that mediate treatment responses, some of which may be modifiable (eg environmental exposures, viruses, disease phenotypes).

The Mount Sinai Therapeutic Infusion Center is an ideal location where investigators have the potential to fill in many of these research gaps. The volume is large, with currently 1803 individuals actively (in 2019) receiving anti-cytokine or anti-CD20 biological treatment for their immunological, dermatological and neurological disorders, largely prescribed by members of the Divisions of Clinical Immunology, Rheumatology, Pulmonary, Inflammatory Bowel Disease (IBD), Neurology and Dermatology. Further, investigators across Divisions (Clinical Immunology, Rheumatology, IBD) and Departments (Medicine, Neurology, Dermatology) have created a research working group to discuss collaborations and standardized approaches to assessing immunological responses to biologics. This registry also intends to coordinate with other registries at ISMMS to ensure that it utilizes common approaches to biomonitoring and common data elements as much as feasible to facilitate comparisons across cohorts.

Primary and Secondary Study Endpoints

The initial scientific hypotheses focus on these endpoints:

Aim 1 An expanded repository of biological specimens and questionnaire data.

Aim 2 Measures of IgE phenotypes and associated clinical airway outcomes.

Aim 3 Measures of changes in the dopaminergic pathway and clinical airway outcomes.

Aim 4 Measures of anti-TNF, anti-CD20, and other biologic therapies on immunological and clinical outcomes.

Aim 5 Measures of IVIG-induced immunological and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years and up.
* Able to provide informed consent.
* Medical care at Mount Sinai.
* Receiving a biologic medication or immune modulator at Mount Sinai, or considered an appropriate negative control or comparison participant by the study team.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing treatment at Mount Sinai Therapeutic Infusion Center will be one major source of participants. Active recruitment will focus on patients new to the Infusion Center. These patients and potential subjects will be densified 1-2 weeks in advance following review of the electronic medical record's schedule by a research study coordinator or other investigator. The primary or referring clinical team, or the current Infusion Center medical team, will let the patient know that a study is available, and if the patient is agreeable, that the research team will contact them.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Biologics and Clinical Immunology Registry | 3 years
  Establish a bioregistry of patients receiving biologic therapy as part of their standard treatment at the Mount Sinai Therapeutic Infusion Center and affiliated practices. The approach is twofold. The first component is to establish a robust and flexible biorepository and database that includes demographic, immunologic, exposure and clinical records, and can facilitate research across disciplines, and across other registries affiliated with Mount Sinai. The second component is to address specific key research questions focused on using novel diagnostics to increase the effectiveness of biologic treatment.

SECONDARY OUTCOMES:
Asthma Control Questionnaire (ACQ) | Up to 3 years
  For patients with asthma. The Asthma Control Questionnaire (ACQ) assess asthma beliefs about asthma control. The ACQ is a 7-item instrument, full scale from 0-6, higher score indicates more impairment.
Multidimensional Health Assessment Questionnaire (MDHAQ) | Up to 3 years
  For patients with rheumatological disorders. Full scale from 0-3, higher score indicates poorer health outcomes.
Clinical Disease Activity Index CDAI) - need information | Up to 3 years
  For patients with rheumatologically disorders who are recruited initially in their rheumatology physician office. Full scale from 0 to 76, with higher score indicating poorer health outcomes.
Birmingham Vasculitis Activity Score (BVA) | Up to 3 years
  For patients with vasculitis. Full scale from 0 to 63, with higher score indicating poorer health outcomes.
Bath Ankylosing Spondylitis Disease Activity | Up to 3 years
  For patients with ankylosing spondylitis. Full scale from 0 to 10, with higher score indicating poorer health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Miller, Principal Investigator — Icahn School of Medicine
Locations (1):
- Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. To achieve aims in the approved proposal. Proposals should be directed to rachel.miller2@mssn.edu. To gain access, data requestors will need to sign a data access agreement.